CLINICAL TRIAL: NCT00290381
Title: The Effects of OC000459 on Nasal Th2 Cytokine Release, Eosinophil Responses, and Nasal Symptoms After Nasal Allergen Challenge (NAC) With Timothy Grass Pollen in Subjects With Allergic Rhinitis Out of Season
Brief Title: The Effects of OC000459 on Nasal Mediators
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Trevor Hansel (Other)
Collaborators: Oxagen Ltd (Industry)
Responsible Party: Sponsor-Investigator, Trevor Hansel, Imperial College, Imperial College London
Organization: Imperial College London (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: OC000459/005/05
Record Dates: First submitted 2006-02-10; First posted 2006-02-13 (Estimated); Last update posted 2023-10-30 (Actual); Status verified 2023-10

CONDITIONS: Allergic Rhinitis
Keywords: Allergic rhinitis
MeSH Terms: conditions — Rhinitis, Allergic

STUDY DESIGN:
Intervention Model Description: Nasal Allergen Challenge Study
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo followed by Drug (OC000459) (Experimental): Placebo and Drug are followed by Nasal Allergen Challenge
  Interventions: Procedure: Oxagen OC000459
- Drug (OC000459) followed by Placebo (Experimental): Drug and Placebo are followed by Nasal Allergen Challenge
  Interventions: Procedure: Oxagen OC000459

INTERVENTIONS:
Procedure: Oxagen OC000459

SUMMARY:
This is the first proof of concept study for OC000459 and is undertaken to assess the effects of the compound on the development of inflammatory cytokines in a model (nasal allergen challenge model) that is validated and clinically safe and easy to conduct. OC000459 will be compared with placebo in the study.

The study will be a randomised, double blind, placebo controlled, crossover evaluation of the effect of OC000459 on cytokine secretion induced by nasal allergen challenge. Male subjects with a known history of allergic rhinitis and screening positive to allergen will be included. After dosing with OC000459 or placebo, nasal allergen challenge will be performed and measurements made in the nasal fluids. Nasal symptom scores will also be recorded. Safety parameters will be monitored throughout.

ELIGIBILITY:
Inclusion Criteria:

1. Males aged 18 to 50 years with a history of symptoms of grass pollen related allergic rhinitis within the previous two years.

Exclusion Criteria:

1. Medical conditions likely to affect the outcome of the study.

2 History of immunotherapy in the past 3 years or currently on an immunotherapy treatment course including inhaled or local corticosteroids in the past 28 days.

3. Any infirmity, disability, or geographic location which, in the opinion of the principal investigator, would limit compliance with the protocol.

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Primary Completion 2005-02-01 (Actual)

PRIMARY OUTCOMES:
The Effect of OC000459 on Nasal Filter Paper Levels of IL-4, IL-5, IL-13 | 1 to 9 hours after nasal allergen challenge

CONTACTS AND LOCATIONS:
Overall Officials: Trevor T Hansel, FRCPath, Principal Investigator — National Heart & Lung Institute
Locations (1):
- National Heart & Lung Institute Clinical Studies Unit, London, United Kingdom

DOCUMENTS (1):
  • Study Protocol (2005-12-22): https://cdn.clinicaltrials.gov/large-docs/81/NCT00290381/Prot_000.pdf